CLINICAL TRIAL: NCT00215982
Title: A Phase II Study of Capecitabine in Combination With Irinotecan and Oxaliplatin (Eloxatin) in Adult Patients With Advanced Colorectal Cancer
Brief Title: Study of Capecitabine With Irinotecan and Oxaliplatin (Eloxatin) in Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Christopher Garrett, M.D., M.D. Anderson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13424; XEL351 (Other: Roche)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Cancer
Keywords: advanced; colon; rectal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Therapy (Experimental): Capecitabine in Combination with Irinotecan and Oxaliplatin
  Interventions: Drug: capecitabine; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: capecitabine — Capecitabine will be administered at a dose of 825 mg/m2 PO BID, for a total daily dose of 1650 mg/m2. Capecitabine will be administered on days 1-14 followed by 7 day treatment free rest period and days 21-35 followed by a 7 day treatment-free rest period, every six weeks (42 days) of treatment is considered one cycle.
  Other Names: XELODA™
Drug: Oxaliplatin — Oxaliplatin will be administered at a dose of 130 mg/m2 IV over 120 minutes in 250-500 ML D5W on day 1, every 42 days.
  Other Names: E LOXATIN™
Drug: Irinotecan — Irinotecan will be administered at a dose of 180mg/m2 IV over 90 minutes on day 21 every 42 days.
  Other Names: CAMPTOSAR™

SUMMARY:
The purpose of this study is to find out how effective the new combination of the drugs Capecitabine (Xeloda), Oxaliplatin (Eloxatin), and Irinotecan (Camptosar) are against colon and rectal cancer. All three of these drugs are approved by the Food and Drug Administration (FDA) for the treatment of colon or rectal cancer. This however is the first time that these three drugs have been combined in this schedule for the treatment of colon/rectal cancer.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the radiographic response rate in patients with metastatic colorectal cancer treated with Oxaliplatin, Capecitabine and Irinotecan. Secondary objectives are to determine the time to tumor progression and the toxicity and tolerability of Oxaliplatin, Capecitabine and Irinotecan when administered in combination. Study schema is as follows. Cycles are 42 days long. Patients will receive Oxaliplatin and Capecitabine on day 1. Capecitabine is an oral pill that will be taken for 14 days. Patients return again on day 21 when they receive Irinotecan and Capecitabine. Capecitabine again is taken for 14 days. CT scans are performed at the end of the 6 week cycle to determine response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmed metastatic colorectal cancer.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* No prior chemotherapy in the metastatic setting (prior fluorouracil chemotherapy, if administered in the adjuvant setting, and if more than 6 months has passed since the completion of therapy, is allowable). Prior adjuvant radiation therapy allowable provided no greater than 30% total bone marrow included in the field (must be more than 6 weeks since completion of radiation therapy.
* Subject must be 18 years or older
* Life expectancy greater than 12 weeks.
* ECOG performance status <2 (Karnofsky >60%).
* Patients must have normal organ and marrow function as defined as: leukocytes >3,000/mcL; absolute neutrophil count >1,500/mcL; Platelets >100,000/mcL; total bilirubin within normal institutional limits; AST(SGOT)/ALT (SGPT) <2.5 X institutional upper limit of normal; Creatinine within normal institutional limits and Creatinine clearance (estimated by Cockcroft-Gault equation)>50-mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of therapy (female patients of childbearing potential).
* Woman of childbearing potential with either a positive or no pregnancy test at baseline. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients will agree to continue contraception for 30 days from the date of the last study drug administration
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior therapy for MCRC in the metastatic setting.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Grade 2 or greater peripheral neuropathy.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Pregnant and nursing women are excluded from this study. Women / men of childbearing potential not using a reliable and appropriate contraceptive method.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with Oxaliplatin and Irinotecan or other agents administered during the study.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* History of clinically significant interstitial lung disease and/or pulmonary fibrosis.
* History of persistent neurosensory disorder including but not limited to peripheral neuropathy
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Any prior platinum based therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
response rate | average of 12 months
  To determine the radiographic response rate in patients with metastatic colorectal cancer treated with Oxaliplatin, Capecitabine and Irinotecan

SECONDARY OUTCOMES:
time to tumor progression | average of 12 months
  To determine the time to tumor progression in patients with metastatic colorectal cancer treated with Oxaliplatin, Capecitabine and Irinotecan
toxicity and tolerability | average of 12 months
  To determine the toxicity and tolerability of Oxaliplatin, Capecitabine and Irinotecan when administered in combination

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Garrett, MD, Principal Investigator — H. Lee Moffitt Cancer Center & Research Institute (now at M.D. Anderson)
Locations (2):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States
- San Juan Veterans Hospital, Rio Piedras, Puerto Rico